CLINICAL TRIAL: NCT01276262
Title: A Single-blind, Placebo-controlled, 2-period, Fixed Sequence Study to Determine the Effects of Coadministration of Fostamatinib 100 mg Twice Daily on the Pharmacokinetics of an Oral Contraceptive in Healthy Female Subjects
Brief Title: Effects of Administration of Fostamatinib on Blood Concentrations of an Oral Contraceptive in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: D4300C00012
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Scientific Terminology Rheumatoid Arthritis, Healthy Female Volunteers, Pharmacokinetics, Oral Contraceptive, Drug-drug Interaction; Laymen Terminology Level of Oral Contraceptive in Blood, Oral Contraceptive, Rheumatoid Arthritis, Drug -Drug Interaction
Keywords: Phase 1, healthy female volunteers, oral contraceptive, pharmacokinetics, Rheumatoid arthritis, RA, fostamatinib
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib; Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Treatment A (Placebo Comparator): Monophasic oral contraceptive (Microgynon® 30) with placebo tablets
  Interventions: Drug: Microgynon® 30 (Oral contraceptive); Drug: Placebo
- Treatment B (Experimental): Monophasic oral contraceptive (Microgynon® 30) and fostamatinib
  Interventions: Drug: fostamatinib; Drug: Microgynon® 30 (Oral contraceptive)

INTERVENTIONS:
Drug: fostamatinib — Oral tablets, repeated doses for 21 days (2 x 50mg BID)
  Arms: Treatment B
Drug: Microgynon® 30 (Oral contraceptive) — Oral tablets, repeated doses
Drug: Placebo — Oral tablets BID, repeated doses for 21 days
  Arms: Treatment A

SUMMARY:
A crossover study to assess the effect of repeated doses of fostamatinib on the levels of oral contraceptive (Microgynon® 30) in the blood of healthy female subjects. The study will consist of a screening period of up to 35 days, followed by 2 treatment periods (28 days each) of an oral contraceptive (Microgynon® 30) in the absence and presence of fostamatinib. The study will also evaluate the safety and tolerability of fostamatinib in combination with an oral contraceptive

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of age 18 to 45 years, inclusive, who are healthy, non-pregnant, not planning pregnancy within the study period
* Willing to use a highly effective method of birth control, ie, double barrier method contraception (condom and diaphragm with spermicide) from the first day of Period 1 until 28 days after the last dose
* Body weight of at least 50 kg and body mass index (BMI) between 18 and 30 kg/m2 inclusive
* Two negative pregnancy tests at least 7 days apart

Exclusion Criteria:

* History of any clinically significant disease or disorder
* History or presence of Gastrointestinal, hepatic, or renal disease
* Any condition listed as a contraindication in the Microgynon® 30 labelling
* Absolute neutrophil count less than 2.5 x 109/L.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To assess the effects of repeated doses of Fostamatinib on the pharmacokinetics of Microgynon ®30 by assessment of Cssmax and AUCss of ethinyl estradiol (EE), levonorgestrel on Day 21 | From predose until Day 22 of each Treatment period

SECONDARY OUTCOMES:
To characterise the PD of progesterone, LH, FSH, and SHBG, following dosing with monophasic oral contraceptive (Microgynon® 30) alone and following coadministration with fostamatinib | From predose until Day 22 of each Treatment period
  PD = pharmacodynamics, LH = luteinising hormone, FSH = follicle stimulating, SHBG = Sex hormone binding globulin
To determine R-406 plasma concentration-time profile and resulting PK parameters including AUCss, Cssmax, and tmaxss | From pre-dose until 12 hours following final dose on Day 21
To determine the safety and tolerability of fostamatinib in combination with an oral contraceptive (Microgynon ®30): adverse event monitoring, vital signs, physical examinations, clinical laboratory tests, ECGs | Screening, treatment periods 1 and 2, Follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, London, United Kingdom